CLINICAL TRIAL: NCT00640211
Title: A Prospective Study to Examine the Effectiveness and Safety of Neuraminidase Inhibitors in Volunteers Who Receive Long-term Prophylaxis Against Pandemic Influenza: PIPET B
Acronym: PIPET B
Status: Withdrawn | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Associate Professor Sean Emery, Therapeutic and Vaccine Research Programme, National Centre in HIV Epidemiology and Clinical Research, University of New South Wales
Other Study IDs: PIPET B
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Pandemic Influenza
Keywords: Prophylaxis; pandemic influenza; influenza A; H5N1 virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PIPET B: Participants in this study will be health care and other essential workers receiving long term neuraminidase inhibitor prophylaxis.

SUMMARY:
This aim of this project is to evaluate the efficacy of neuraminidase inhibitors as prophylaxis against pandemic influenza infection in patients who are prescribed a long term course in the context of a place of employment or profession. The study is observational only. The primary measure used in this study will be the incidence of symptomatic pandemic influenza in patients receiving prophylaxis. Seroconversion to pandemic influenza, the incidence of adverse events and the relative effectiveness of oseltamivir and zanamivir prophylaxis will also be examined. This project will commence upon pandemic influenza being declared in Australia, Hong Kong or Singapore. Data will be analysed as quickly as possible to help inform the continued use of neuraminidase inhibitor therapy as a cornerstone of the public health agency response to pandemic influenza.

DETAILED DESCRIPTION:
The aim of this study is to

1. Describe the incidence of symptomatic pandemic influenza infection in participants receiving neuraminidase inhibitor prophylaxis in the context of a place of employment or a profession
2. Describe the incidence of seroconversion to pandemic influenza
3. Describe the incidence of adverse events in volunteers taking long term antiviral prophylaxis
4. Compare the effectiveness of oseltamivir and zanamivir prophylaxis

The study is an open label prospective cohort study. Participants in this study will be health care and other essential workers receiving long term neuraminidase inhibitor prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Intention to commence, or already commenced prophylaxis with a neuraminidase inhibitor in the context of a place of employment or profession

It is anticipated that participants in this study who are subsequently clinically diagnosed with pandemic influenza will be enrolled in the Index Case protocol (PIPET-A) with follow-up as specified.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study will be health care and other essential workers receiving long term neuraminidase inhibitor prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The primary measure used in this study will be the incidence of symptomatic pandemic influenza in patients receiving prophylaxis. | One month

SECONDARY OUTCOMES:
Seroconversion to pandemic influenza, the incidence of adverse events and the relative effectiveness of oseltamivir and zanamivir prophylaxis will also be examined. | One month

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Dwyer, Principal Investigator — Westmead Hospital
Locations (8):
- Australia (8):
  - St Vincent's Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia